CLINICAL TRIAL: NCT04363411
Title: Reaching Out to the UNdiagnosed People Infected With Blood Borne Viral Infections
Acronym: RUNtoBBV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Geert Robaeys, Principal Investigator, Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RUNtoBBV-001
Record Dates: First submitted 2020-01-07; First posted 2020-04-27 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Hepatitis B; Hepatitis c; Human Immunodeficiency Virus
MeSH Terms: conditions — Hepatitis B; Hepatitis C; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- drug use (Experimental)
  Interventions: Other: finger prick screening for BBV infections and questionnaires by outreaching methodology

INTERVENTIONS:
Other: finger prick screening for BBV infections and questionnaires by outreaching methodology — Screening by fingerprick for HCV Ab, HBsAg and HIV Ab and a questionnaire will be performed at sites outside of the regular treatment facilities.

SUMMARY:
Title Reaching out to the UNdiagnosed people infected with blood-borne viral infections (RUNtoBBV) Objectives 1. To study the efficacy of an outreach methodology to increase the uptake for screening, linkage to care and treatment in (active or former) people who use drugs (PWUD) Trial design Prospective multicenter interventional cohort design Number of subjects 336 inclusions (with prevalence of HCV Ab: 30%)

* 168 Antwerp
* 168 Limburg

Selection criteria Inclusion criteria:

* 18 years of age
* History of/ or active drug use
* Written informed consent obtained Exclusion criteria
* Currently enrolled in centralized OST program of Free Clinic or CAD Limburg Endpoints The following endpoints will be compared between the centers in Limburg and Antwerp: (Main outcome in bold)

Main objectives:

* Prevalence of blood-borne viral infections in Belgian (former or active) PWUD:

  * HCV infection (number of HCV Ab+ / number of screened PWUD)
  * HBV infection (number of HBsAg+/number of screened PWUD)
  * HIV infection (number of HIV Ab+/number of screened PWUD)
* Analysis of linkage to care to hepatologist/ infectiologist (number of patients who adhered to their consultation/number of referred patients)

Secondary objectives:

* Analysis of risk behavior/sociodemographics linked to presence of BBV infections
* Analysis of uptake of anti(retro)viral treatment (number of patients started on treatment/number of patients needing treatment)
* Analysis of treatment adherence (adherence to treatment consultations/total planned consultations)
* Analysis of treatment outcome (total number of cured or virally suppressed patients/total number of treated patients)

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* History of drug use
* Active drug use
* Written informed consent obtained

Exclusion Criteria:

* Currently enrolled in OST program of Free Clinic or CAD Limburg (centralized OST provision)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2019-10-22 (Actual)

PRIMARY OUTCOMES:
HCV Ab+ (Hepatitis C Virus antibody) | day 1
  test using whole capillary blood (finger prick testing)
HBsAg+ (Hepatitis B surface Antigen) | day 1
  test using whole capillary blood (finger prick testing)
HIV Ab+ (human immunodeficiency virus) antibody | day 1
  test using whole capillary blood (finger prick testing)

SECONDARY OUTCOMES:
4. Questionnaire to Identify risk factors associated with the aforementioned blood borne viral infections (hepatitis C, hepatitis B and HIV) | day 1
  i. Combine results from positive finger prick test with questionnaire regarding sociodemographic factors, migration, risk factors for blood born viruses (sexual contacts, incarceration, drug use). The questionaire does not include a score on scale.
Analysis of uptake of anti(retro)viral treatment | Day 1
  percentage of HCV positive clients who started treatment in relation of total of HCV positive clients needing treatment
Analysis of treatment adherence | up to one year
  percentage of patients reaching end-of treatment response, who present at the consultation, in relation to total patients in treatment
Analysis of treatment outcome | month 18
  total number of cured or virally suppressed patients/total number of treated patients

CONTACTS AND LOCATIONS:
Overall Officials: Geert Robaeys, prof. dr., Principal Investigator — Hasselt University; Rob Bielen, dr., Study Chair — Hasselt University
Locations (10):
- Belgium (10):
  - Free Clinic Antwerpen, Antwerp
  - Free Clinic Antwerp, Antwerp
  - ZNA Antwerp, Antwerp
  - Ziekenhuis Oost-Limburg, Genk
  - CAD Limburg, Hasselt
  - Jessa Ziekenhuis, Hasselt
  - Ziekenhuis Maas en Kempen, Maaseik
  - Mariaziekenhuis Noord-limburg, Overpelt
  - AZ Sint-Trudo, Sint-Truiden
  - AZ Vesalius, Tongeren

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Busschots D, Kremer C, Bielen R, Koc OM, Heyens L, Dercon E, Verrando R, Windelinckx T, Maertens G, Bourgeois S, Hens N, Mathei C, Robaeys G. Identification and treatment of viral hepatitis C in persons who use drugs: a prospective, multicenter outreach study in Flanders, Belgium. Harm Reduct J. 2021 May 17;18(1):54. doi: 10.1186/s12954-021-00502-7. PMID 34001145